CLINICAL TRIAL: NCT01176877
Title: Assessing and Improving Patient Knowledge About Keloids
Brief Title: Assessing and Improving Patient Knowledge About Keloid Scars (Keloids)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Roopal Kundu, Associate Professor of Dermatology, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: STU32316
Record Dates: First submitted 2010-07-30; First posted 2010-08-06 (Estimated); Results first posted 2013-01-03 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-11

CONDITIONS: Keloid Scar
MeSH Terms: conditions — Keloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- keloid scar (Other): Those with a diagnosis of keloid scar.
  Interventions: Behavioral: Scripted lecture ("educational information talk")

INTERVENTIONS:
Behavioral: Scripted lecture ("educational information talk") — This scripted lecture will be approximately 5 minutes in length and will include 3 picture examples of keloid and hypertrophic scarring as well as an opportunity to ask questions.

SUMMARY:
The purpose of this study is:

* to identify how knowledge about keloid scars and self-treatments differs between patients who use the Internet as a source of information and patients who do not
* to determine if patients who are at a high risk of developing additional keloid scars are more or less likely to change their behavior based on an educational information talk about keloid scar prevention

DETAILED DESCRIPTION:
Keloids scars differ from other scar types in that they grow beyond the borders of the injury that caused them. Patients with darker pigmented skin are more likely to develop keloids, and blacks are especially predisposed to keloid formation. Treatment options for keloids are limited in that new keloids often form at the treated location. The limited efficacy of professional treatment options and the harmless appearance of small keloid scars may lead a patient to try to manage their keloid scars on their own. One source of information that patients may turn to for self-treatment advice is the Internet.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a clinical diagnosis of keloid scarring
* Subjects over the age of 18

Exclusion Criteria:

* That which does not fit the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roopal V Kundu, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States

REFERENCES:
- [Background] Juckett G, Hartman-Adams H. Management of keloids and hypertrophic scars. Am Fam Physician. 2009 Aug 1;80(3):253-60. PMID 19621835
- [Background] Sclafani AP, Gordon L, Chadha M, Romo T 3rd. Prevention of earlobe keloid recurrence with postoperative corticosteroid injections versus radiation therapy: a randomized, prospective study and review of the literature. Dermatol Surg. 1996 Jun;22(6):569-74. doi: 10.1111/j.1524-4725.1996.tb00376.x. PMID 8646474
- [Background] Shaffer JJ, Taylor SC, Cook-Bolden F. Keloidal scars: a review with a critical look at therapeutic options. J Am Acad Dermatol. 2002 Feb;46(2 Suppl Understanding):S63-97. doi: 10.1067/mjd.2002.120788. PMID 11807470
- [Background] Shinchuk LM, Chiou P, Czarnowski V, Meleger AL. Demographics and attitudes of chronic-pain patients who seek online pain-related medical information: implications for healthcare providers. Am J Phys Med Rehabil. 2010 Feb;89(2):141-6. doi: 10.1097/PHM.0b013e3181c56938. PMID 19966558
- See also: Northwestern University Department of Dermatology Actively Enrolling Research Trials — http://www.feinberg.northwestern.edu/depts/dermatology/research/clinical-trials/ctu-active%20trials.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between August 2010 and June 2011, 40 subjects were recruited from patients seen for keloid scars at Northwestern University's dermatology clinic in Chicago, Illinois, and from the general population by advertisements in a local newspaper and Internet classified ads.
Groups:
- Keloid Scar: Subjects over the age of 18 with a clinical diagnosis of keloid scarring were included in the study. First, subjects completed a written questionnaire to collect demographic data, including personal history of keloid scarring, past and present use of keloid scar treatments, and internet access and use to find information related to keloid scars. Second, subjects completed a written questionnaire to assess knowledge about keloids. Next, subjects listened to a scripted, 5 minute educational lecture about keloid scars and then completed a written questionnaire to assess knowledge about keloids. Finally, subjects were contacted by phone 3 months later to complete a questionnaire to assess knowledge about keloids and to answer questions about keloid-related behaviors over the previous 3 months.
Period: Overall Study
Arm/Group | Keloid Scar
Started | 40
Completed | 31
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Keloid Scar
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 2
Age Continuous [Mean (Inter-Quartile Range); unit: years] | 40 [29 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Impact of an Educational Lecture on Knowledge About Keloid Scars by Comparing Mean Scores Between Knowledge Assessment Questionnaires Administered Before an Educational Lecture and Immediately After an Educational Lecture
Description: All subjects completed a written questionnaire to assess knowledge about keloid scars before an educational lecture about keloids, immediately after the educational lecture about keloids, and 3 months after the educational lecture about keloids. This written questionnaire to assess knowledge about keloid scars contained 19 questions related to risk factors for developing keloid scars, keloid scar prevention, and keloid scar treatment. A correct response to a question was awarded 1 point and all correct responses were summed to achieve a total score. Possible total score ranged from 0 to 19. A score of 0 is associated with worse knowledge about keloid scars and a score of 19 is associated with better knowledge about keloid scars.
Time Frame: immediately before and after a 5 minute educational lecture
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Keloid Scar: Participants with keloid scars completed a written questionnaire to assess knowledge about keloid scars. Participants then listened to a scripted, 5 minute educational lecture about keloid scars. Immediately after the educational lecture, the subjects completed an identical written questionnaire to assess knowledge about keloid scars.
Arm/Group | Keloid Scar
Number analyzed (Participants) | 40
score on a scale
  Pre-educational lecture score | 12.9 [5 to 19]
  Immediate post-educational lecture score | 18.3 [14 to 19]

2. Secondary Outcome: To Assess the Impact of an Educational Lecture on Long-term Knowledge Retention About Keloid Scars by Comparing Mean Scores Between Knowledge Assessment Questionnaires Administered Before an Educational Lecture and 3 Months After an Educational Lecture
Description: as for outcome 1
Time Frame: before and 3 months after a 5 minute educational lecture
Population: Patients enrolled who were available for phone contact 3 months following intervention.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Keloid Scars: Participants with keloid scars completed a written questionnaire to assess knowledge about keloid scars. Participants then listened to a scripted, 5 minute educational lecture about keloid scars. 3 months after the educational lecture, subjects completed an identical verbal questionnaire to assess knowledge about keloid scars.
Arm/Group | Keloid Scars
Number analyzed (Participants) | 31
score on a scale
  Pre-educational lecture score | 13.2 [5 to 19]
  3 months post-educational lecture score | 16.8 [12 to 19]

ADVERSE EVENTS:
Arm/Group | Keloid Scar
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

LIMITATIONS AND CAVEATS:
limitation of the study is the accrual of a majority of participants from keloid patients at a single academic center.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes